CLINICAL TRIAL: NCT01198717
Title: Multicentre Paediatric Disease Registry in Essential Thrombocythaemia
Brief Title: Pediatric Disease Registry in Essential Thrombocythaemia (ET)
Status: Completed | Type: Observational
Sponsor: Shire (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Other Study IDs: SPD422-404
Record Dates: First submitted 2010-09-08; First posted 2010-09-10 (Estimated); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Essential Thrombocythemia (ET)
MeSH Terms: conditions — Thrombocythemia, Essential

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this study is to evaluate the progression of ET in children (aged 6-17years inclusive) over a period of 5 years maximum. The study will also assess how children are diagnosed, treatment options for those children with symptoms and events related to their ET and the outcomes of those treatments.

ELIGIBILITY:
Inclusion Criteria:

- 6 years or over and less than 18 years patient has ET according to the WHO criteria as guidance

Exclusion Criteria:

* Interventional clinical study participation

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Paediatrics aged between 6 years and 17 years
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2010-09-28 (Actual); Primary Completion 2016-03-01 (Actual); Study Completion 2016-03-01 (Actual)

PRIMARY OUTCOMES:
Treatment effects on platelet count in children ages 6-17 years inclusive. | 60 months

SECONDARY OUTCOMES:
Drug utilization of cytoreductive therapy in children ages 6-17 years inclusive | 60 months

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (32):
- Czechia (2):
  - Paediatric Clinic University Hospital Olomouc, Olomouc
  - Clinic of Paediatric haematology and oncology University Hospital Motol, Prague
- France (4):
  - Paediatric Oncology Unit, Hopital Cote De Nacre, Caen
  - Practicen Hospitalier , Institute d'Hematologie et Oncologie Pediatrique, Lyon
  - Centre Hospitalier Lyon Sud - service Hématologie, Pierre-Bénite
  - Hopitaux de Brabois, Vandœuvre-lès-Nancy
- Germany (2):
  - Klinikum Chemnitz GmbH, Klinik für Kinder-und Jugendmedizin, Chemnitz
  - Zentrum für Kinder- und Jugendmedizin Klinik II / III, Frankfurt
- "Agia Sophia" Children's Hospital, Athens, Greece
- Italy (10):
  - Dipartimento di Biomedicina dell'Eta Evolutiva. University of Bari, Bari
  - Servico de Oncoematologia Peditrica, Cagliari
  - UO Oncoematologia AOU Meyer, Florence
  - Pediatric Hamatology Unit. Department of Hematology and Oncology. G Gaslini Children's hospital. Largo, Genova
  - Chairmen of Pediatric Hamatooncology Outpatient Clinic. Hospital San Gerardo, Monza
  - Department of Oncology, Pausilipon Hospital, AORN Santobono, Napoli
  - Azienda Ospedaliera di Padova, Padua
  - Department of Cellular Biotechnologies and Hematology. Sapienza University, Rome
  - Ospedale Casa Sollievo della Sofferenza, San Giovanni
  - Hamatology Unit. Paediatric Department. University of Torino, Torino
- Spain (8):
  - Sección de Hematología Pediátrica. Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Mutua de Terrassa, Barcelona
  - Jefe de Servicio Oncología Y Hematología Pediátricas, Barcelona
  - Servicio de Hematología Clínica, Hospital Sant Joan de Déu Barcelona, Barcelona
  - Servicio de Transfusión, Hospital Universitario Niño Jesús, Madrid
  - Department Haematology, Hospital Ramon y Caja, Madrid
  - Hospital Universitario Virgen de la Arrixac, Murcia
  - Complexo Hospitalario Universitario, Santiago, Santiago de Compostela
- Leitender Arzt, Pädiatrische Hämatologie/Onkologie Kinderspital, Lucerne, Switzerland
- United Kingdom (4):
  - St James University Hospital, Leeds
  - Royal Manchester Childrens Hospital,, Manchester
  - Children's Clinic, Royal Berkshire Hospital, Reading
  - Sheffield Childrens Hospital, Sheffield

REFERENCES:
- See also: To obtain more information on the study, click here/on this link. — https://clinicaltrials.takeda.com/study-detail/5f6b5fee4db2bf003ab47e5c